CLINICAL TRIAL: NCT05040191
Title: The Effect of Haptic Interactive Virtual Reality and Computer-Based Simulation Technologies on Students' Achievement and Anxiety Levels in Nasogastric Tube Practice Teaching
Brief Title: The Effect of Haptic Interactive Virtual Reality on Nasogastric Tube Practice Teaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Hamiyet KIZIL, RN Msc Lecturer, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1870
Record Dates: First submitted 2021-08-17; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Simulation; Nasogastric Tube
Keywords: virtual reality; simulation; nasogastric tube; haptic glove

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Experimental): Application in the Control Group: After the theoretical lesson, the control group was taken to the Nursing Fundamentals Skills Laboratory. The laboratory consists of 3 practice rooms, 1 control room and 1 analysis room. A video prepared by the researcher on the Simple Nasogastric Tube Application Model in line with the steps of "Checklist for Teaching Nasogastric Tube Application Skills" was watched and preliminary information was given. The questions were answered by allowing the students to ask questions.
  Interventions: Other: Traditional Education(control)
- Haptic Interactive Virtual Reality Simulation(Experiment 1 group) (Experimental): Application in the Experiment-1 Group: After the theoretical lesson, the students in the Experiment-1 group were taken to the computer laboratory room where the haptic interactive virtual reality application was installed. The Nasogastric Tube Application with Haptic Interactive Virtual Reality Simulation was applied and explained by the researcher and preliminary information was given. The questions were answered by allowing the students to ask questions.
  Interventions: Other: Haptic interactive virtual reality simulation training
- Haptic Interactive Computer Based Simulation(Experiment 2 group) (Experimental): Application in the Experiment-2 Group: After the theoretical lesson, the students in the Experiment-2 group were taken to the laboratory room where the haptic interactive computer-based simulation was located. This computer-assisted simulation allows us to see the application on the computer screen while performing an application with a haptic arm. It gives feedback on hand manipulations similar to reality. It was explained by the researcher by applying the nasogastric tube application skill with haptic interactive computer-based simulation and preliminary information was given. The questions were answered by allowing the students to ask questions.
  Interventions: Other: Haptic interactive computer-based simulation training

INTERVENTIONS:
Other: Traditional Education(control) — The application was made on the model that allows nasogastric tube application and the anatomical structure in the nasogastric region is seen. The student can experience the skill of applying a nasogastric tube to the nasogastric or orgastric region on this model. In the nursing skills laboratory, students were given a demonstration of nasogastric tube application on a model.
  Arms: Control Group
Other: Haptic interactive virtual reality simulation training — Haptic interactive virtual reality simulation technology; It functions by using haptic gloves that are interactive, visually enhanced, containing three-dimensional video and animation, wearable by students. This program has been developed by a software developer who is an expert in the field of information technologies, using the unreal program with a nine-generation computer with a game engine. All the necessary steps in the NGT application have been in simulation.
  Arms: Haptic Interactive Virtual Reality Simulation(Experiment 1 group)
Other: Haptic interactive computer-based simulation training — "Clinical tvr (tactile simulator)" produced by a foreign commercial company used in nursing education was used. Clinical tvr simulation applications can be accessed online or downloaded to a computer. This simulator; It functions by using an interactive, visually enhanced 2D, animated, haptic arm that can be held by students like a pen. It includes applications such as nasogastric tube placement, urinary bladder catheter placement, heart massage. These applications can be realized through both mouse and haptic arm computer input devices. clinical tvr; It is a simulator that incorporates the enhanced benefits of haptic feedback through the use of haptic technology. This simulator provides a near-realistic sensory experience where the learner can practice a skill as it actually is. Computer-based simulation with haptic interaction was used in this study with the haptic arm in NGT application skill.
  Arms: Haptic Interactive Computer Based Simulation(Experiment 2 group)

SUMMARY:
This research was carried out as a randomized controlled experimental study to evaluate the effects of haptic interactive virtual reality and computer-based simulation technologies on students' knowledge, skills, anxiety, satisfaction in learning and self-confidence in teaching nasogastric tube application.

The research population consisted of students who enrolled in a foundation university nursing department and took the "Basic Principles and Practices in Nursing II" course in the Spring Semester of the 2020-2021 academic year, and the sample consisted of 90 students who met the inclusion criteria of the study. During nasogastric tube application, the Control Group (n=30) trained with the Standard Curriculum, Experimental Group 1 (n=30) trained with Haptic Interactive Virtual Reality Simulation Technology, and Experimental Group 2 (n=30) trained with Haptic Interactive Computer-Based Simulation. n=30) was performed. Research data were collected with "Structured Student Introduction Form", "Nasogastric Tube Application Skills Examination", "Nasogastric Tube Application Skill Checklist", "State-Trait Anxiety Inventory", "Student Satisfaction and Self-Confidence in Learning Scale". Appropriate statistical methods were used in the analysis of the data.

DETAILED DESCRIPTION:
Traditional learning methods and environments are thought to be insufficient to respond to the differing expectations of generation z, who were born and raised in a digital age. For this reason, it has become mandatory for educational institutions to renew their curricula and support them with advanced technologies. All over the world, higher education programs are trying to expand their educational capacities by applying innovative strategies to meet the future workforce needs. Nursing educators also report that fundamental changes in existing curricula are necessary for innovation. Since nursing is a profession that requires the acquisition of cognitive, psychomotor and attitudinal behaviors, it is important to use innovative practices in education. While these applications increase the attention of the student, they save the education from monotony and ensure the permanence of the education by ensuring the active participation of the student. Due to the fact that today is the age of technology, the use and development of new learning tools has increased at every stage of the nursing education process. These developments in technology and education have brought together these two fields and the use of simulation applications used to increase technical and non-technical skills in nursing education has become widespread.

Nasogastric tube (NGT) application, which is one of the interventions that students should develop in nursing education, is an invasive intervention that is frequently applied for enteral nutrition, drug administration and gastric decompression and is the responsibility of health professionals.

Since the beginning of professional nursing education, different teaching methods have been applied to improve nasogastric tube application skills.

According to traditional teaching methods, in teaching NGT practice skill, educators explain the purpose, indications, complications, application method, necessary materials and nursing interventions that need attention in the classroom. Then, demonstration of NGT application skill on a model is made in order to transform theoretical knowledge into behavior in nursing skills laboratories. Due to the fact that it is an invasive procedure with various complications, NGT application by students in the clinical field is limited, so the development and reinforcement of the behavior is left after graduation. It is envisaged that in the teaching of NGT application skill with haptic interactive virtual reality simulation technology, students' knowledge, skills and self-confidence levels will increase, allowing them to feel like a nurse in the patient room that reflects the real hospital conditions, and they will develop and reinforce the NGT application skill, which is a complex initiative in a risk-free environment before graduation. Based on this information, the aim of this study is to reveal the effects of haptic interactive virtual reality and computer-based simulation technologies on students' knowledge, skills, anxiety, satisfaction in learning and self-confidence in teaching nasogastric tube application.

ELIGIBILITY:
Inclusion Criteria:

Students;

* Over 18 years old,
* Registered in the nursing department,
* Able to use a computer,
* No vision and hearing problems
* Have not done the NGT skill practice before,
* Taking the Nursing Fundamentals course for the first time.

Exclusion Criteria:

Students;

* Under 18 years old,
* Can't use a computer,
* Having vision and hearing problems,
* Have done NGT skill practice before,
* Having taken the Nursing Fundamentals course before.

Ages: 19 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
nasogastric tube application skill success levels | 2 Months
  Students were informed about the "Nasogastric Tube Application Skill Checklist"

SECONDARY OUTCOMES:
Anxiety levels | 2 Months
  Students were informed about the "State-Trait Anxiety Inventory"

OTHER OUTCOMES:
Satisfaction and self-confidence levels | 2 Months
  Students were informed about the "Student Satisfaction and Self-Confidence in Learning Scale"

CONTACTS AND LOCATIONS:
Overall Officials: Hamiyet Kızıl, RN Msc, Principal Investigator — Beykent University Istanbul,Turkey
Locations (1):
- Beykent University, Istanbul, Beykent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] SENDIR, M., & KIZIL, H. (2019). An innovative approach in teaching nasogastric tube application: NAZO-AR. Journal of Duzce University Institute of Health Sciences, 9(2), 86-90.
- [Result] Choi KS, He XJ, Chiang VC, Deng Z, Qin J. A Heuristic Force Model for Haptic Simulation of Nasogastric Tube Insertion Using Fuzzy Logic. IEEE Trans Haptics. 2016 Jul-Sep;9(3):295-310. doi: 10.1109/TOH.2016.2550044. Epub 2016 Apr 6. PMID 27071195